CLINICAL TRIAL: NCT07220551
Title: An Open-Label, Single-Center, Randomized, 2-Way Crossover Study to Evaluate the Relative Bioavailability and Safety of Two UCB0022 Tablet Formulations in Healthy Participants
Brief Title: A Phase 1 Relative Bioavailability Study of UCB0022 Tablets in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: UCB Biopharma SRL (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: UP0159
Record Dates: First submitted 2025-10-22; First posted 2025-10-24 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Healthy Volunteers
Keywords: Healthy Volunteers;; UCB0022;; Glovadalen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment Sequence AB (Experimental): Study participants will receive a single oral dose of UCB0022 Formulation 1 (reference) on Day 1 (dosing day of Period 1) and a single oral dose of UCB0022 Formulation 2 (test) on Day 15 (dosing day of Period 2) in Treatment sequence A-B.
  A washout period of 14 days is included for elimination of the drug between the single oral administrations of UCB0022 in Periods 1 and 2.
  Interventions: Drug: UCB0022
- Treatment Sequence BA (Experimental): Study participants will receive a single oral dose of UCB0022 Formulation 2 (test) on Day 1 (dosing day of Period 1) and a single oral dose of UCB0022 Formulation 1 (reference) on Day 15 (dosing day of Period 2) in Treatment sequence B-A.
  A washout period of 14 days is included for elimination of the drug between the single oral administrations of UCB0022 in Periods 1 and 2.
  Interventions: Drug: UCB0022

INTERVENTIONS:
Drug: UCB0022 — Participants will receive a single oral dose of UCB0022 tablet Formulation 1 and UCB0022 tablet Formulation 2 following a pre-specified sequence.
  Other Names: Glovadalen

SUMMARY:
The purpose of this study is to estimate the relative bioavailability of UCB0022 Formulation 2 (Test) versus Formulation 1 (Reference) in healthy participants following single oral administration.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be minimum 18 years and maximum 55 years of age inclusive at the time of signing the informed consent form (ICF).
* Participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, and cardiac monitoring.
* Participants have a blood pressure (BP) and heart rate (HR) during the Screening Period or before the first dose of study intervention, as determined by triplicate BP/HR measurements in a supine position, of mean systolic BP ranging between 90mmHg and 130mmHg, mean diastolic BP ranging between 50mmHg and 80mmHg, and mean HR between 45bpm and 90bpm.
* Body weight greater than or equal (≥)45 kilograms (kg) and body mass index within the range 18.0 kilograms per meter square (kg/m2) to 30.0 kg/m2 (inclusive).
* A male participant must agree to use contraception during both Periods and for at least 14 days after the final dose of study intervention, and refrain from donating sperm during this period.
* A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least 1 of the following conditions applies:

  * Not a woman of childbearing potential (WOCBP) OR
  * A WOCBP who agrees to follow the contraceptive guidance during both Periods and for at least 14 days after the final dose of study intervention.
* Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the ICF and in the protocol.

Exclusion Criteria:

* Participants have any medical or psychiatric condition that, in the opinion of the investigator, could jeopardize or would compromise the study participant's ability to participate in this study.
* History or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrinological, hematological, cerebrovascular, neurological, or other major disorders capable of significantly altering the absorption, metabolism, or elimination of drugs.
* History of hypertension, hypertensive crisis, hypertensive encephalopathy, or orthostatic hypotension
* History of ischemic stroke, transient ischemic attack, angina, myocardial infarction, any systemic embolism, any clinically significant arrythmia, or congestive heart failure.
* Participants have the following liver enzyme test results during the Screening Period or Day -1:

alanine aminotransferase (ALT), aspartate aminotransferase (AST), bilirubin, or alkaline phosphatase (ALP) >1.0×upper limit of normal (ULN) (isolated bilirubin <1.5×ULN is acceptable if fractionated and direct bilirubin <35%).

* Current or chronic history of liver disease or known hepatic or biliary abnormalities (with the exception of asymptomatic gallstones).
* Participants have 12-lead electrocardiogram (ECG) with changes considered to be clinically significant (eg, QTcF >450ms in males and >470ms in females , left bundle branch block, evidence of myocardial ischemia, or second-degree Type II atrioventricular block).
* Participants have a history of risk factors for torsades de pointes.
* Participants have had any malignancy within the past 5 years except for basal cell or squamous epithelial carcinomas of the skin that have been resected with no evidence of metastatic disease for 3 years.
* Participants have had breast cancer within the past 10 years.
* Participants have a history of severe allergic reaction that required medical intervention.
* Participants have a positive HBsAg, hepatitis C virus antibody, or human immunodeficiency virus 1 and 2 antibody result at the Screening Visit.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2025-10-23 (Actual); Primary Completion 2025-12-16 (Actual); Study Completion 2025-12-16 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration-time curve of UCB0022 | From Day 1 (Predose) up to Day 14 of Period 1 and from Day 15 (Predose) up to Day 28 of Period 2
  AUC: Area under the plasma concentration-time curve.
Area under the plasma concentration-time curve from time 0 to t of UCB0022 | From Day 1 (Predose) up to Day 14 of Period 1 and from Day 15 (Predose) up to Day 28 of Period 2
  AUC0-t: Area under the plasma concentration-time curve from time 0 to t.
Maximum observed plasma concentration of UCB0022 | From Day 1 (Predose) up to Day 14 of Period 1 and from Day 15 (Predose) up to Day 28 of Period 2
  Cmax: Maximum observed plasma concentration.

SECONDARY OUTCOMES:
Occurrence of Treatment-emertgent Adverse Events (TEAEs) from Day 1 up to end of the Safety Follow-up (SFU) Period or End of Study (EOS) | From Dosing (Day 1) up to SFU period or End of study (EOS) (up to Day 28)
  A TEAE is defined as any AE with a start date or time on or after the first dose of study intervention until the end of the SFU Period (ie, EOS/SFU Visit).

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 0018445992273
Locations (1):
- UP0159 1, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No
Due to the small sample size in this trial, individual patient-level data cannot be adequately anonymized i.e., there is a reasonable likelihood that individual participants could be re-identified. For this reason, data from this trial cannot be shared.